CLINICAL TRIAL: NCT01346202
Title: Influence of a Multimodal Day-unit Pain Therapy on Pain Experience, Pain-related Disability and Depression in Patients With Chronic Pain Syndromes
Brief Title: Effects of Multimodal Pain Therapy in Patients With Mixed Chronic Pain Syndromes
Acronym: IMPERApain
Status: Completed | Type: Observational
Sponsor: Klinikum St. Georg gGmbH (Other)
Responsible Party: Principal Investigator, Armin Sablotzki, MD, Prof. Dr. med., Klinikum St. Georg gGmbH
Other Study IDs: EK-BR-28/10-1
Record Dates: First submitted 2011-04-27; First posted 2011-05-02 (Estimated); Last update posted 2013-07-15 (Estimated); Status verified 2013-07

CONDITIONS: Chronic Pain
Keywords: multi-modal pain therapy, chronic pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- chronic pain: 260 consecutive patients with verified chronic pain syndromes

SUMMARY:
Complex and chronified pain syndromes requires a specialized therapeutic concept. From patients with chronic low back pain the investigators know, that an interdisciplinary multi-modal approach may improve the therapeutic success. In this observational study the investigators investigated if the multi-modal pain therapy is also effective in patients with mixed chronic pain syndromes.

DETAILED DESCRIPTION:
The multi-modal pain therapy includes:

* specific drug therapy
* pain education
* psychological therapy
* physical therapy
* behavioral therapy
* work hardening
* bio-feedback
* ergotherapy

ELIGIBILITY:
Inclusion Criteria:

* age >= 18 years and <= 65 years
* verified chronic pain for more than 6 month

Exclusion Criteria:

* application for a pension
* non-accordance with multi-modal pain therapy
* dominant geriatric symptoms
* dominant psychiatric symptoms

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 260 consecutive patients with chronic pain syndromes
Sampling Method: Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2011-01; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
intensity of pain | Change from Baseline in intensity of pain at 1 year
  pain intensity 1 year after multi-modale therapy compared with pain intensity before treatment

SECONDARY OUTCOMES:
pain disability index | Change from Baseline in pain disability index at 6 months
  pain disability index 6 month after multi-modale therapy compared with pain disability index before treatment

CONTACTS AND LOCATIONS:
Overall Officials: Armin R Sablotzki, MD, PhD, Principal Investigator — Klinikum St. Georg
Locations (1):
- Klinikum St. Georg, Pain Center, Leipzig, Saxony, Germany

REFERENCES:
- See also: Related Info — http://www.sanktgeorg.de